CLINICAL TRIAL: NCT02124174
Title: Maintenance Therapy With Azacitidine and Valproic Acid After Allogeneic Stem Cell Transplant in Patients With High-Risk Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS)(Version 1_06 Jan 2012)
Brief Title: Vidaza and Valproic Acid Post Allogeneic Transplant for High Risk AML and MDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Patrick Stiff (Other)
Responsible Party: Sponsor-Investigator, Patrick Stiff, Professor, Loyola University
Organization: Loyola University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203835
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Acute Myelogenous Leukemia AML; Myelodysplastic Syndrome MDS
Keywords: acute myelogenous leukemia (AML); myelodysplastic syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Myelodysplastic Syndromes | interventions — Azacitidine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vidaza and Valproic Acid (Experimental): Vidaza and Valproic Acid
  Interventions: Drug: Vidaza and Valproic Acid

INTERVENTIONS:
Drug: Vidaza and Valproic Acid — Days 1-5: 5-Azacytidine 40 mg/m^2 daily Days 1-5: +Valproic acid 15 mg/kg daily Days 6-28: Valproic acid 15 mg/kg daily
  *treatments will be repeated on the same days of each cycle for up to 4 total cycles. Each cycle will consist of 28 days.
  Other Names: Vidaza; Valproic Acid; Azacitadine

SUMMARY:
Phase II trial combining azacitidine with valproic acid as maintenance therapy post allogeneic stem cell transplantation in patients with high-risk MDS/AML. We hypothesize that adding valproic acid to azacitidine will improve outcomes via both direct anti-tumor and immunologically mediated antitumor response with alloreactive donor lymphocytes, having an additive effect and extending 1 year survival in patient with high-risk AML/MDS after hematopoietic stem cell transplant. Based on aforementioned data from the US Department of Health and Human Services, standard 1 year survival for AML after stem cell transplant is near 40%. We hypothesize that valproic acid and azacitidine will prolong survival, with a 1 year survival goal of 60%. In addition to assessing for 1 year survival, we will have secondary objectives of assessing progression-free survival, relapse, and toxicity. The primary toxicity endpoint from this will be cytopenias and infections.

DETAILED DESCRIPTION:
To assess the combination of valproic acid and azacitidine in preventing relapse in patients with high-risk Acute Myeloid Leukemia (AML) and myelodysplastic syndrome (MDS) after allogeneic stem cell transplant. The primary objective of this study will be determining the 1 year overall survival from combining valproic acid (VPA) with 5-azacytidine (5-aza).

To assess the effect that adding valproic acid to azacitidine will have in patient with high-risk Acute Myeloid Leukemia (AML) and myelodysplastic syndrome (MDS) after allogeneic stem cell transplant on the following endpoints

ELIGIBILITY:
Inclusion Criteria:

1. All allograft patients > 2 years of age.
2. Patients will have one of the following malignancies:

   a. Patients with refractory or relapsed: acute myelogenous leukemia (AML) (including inv16, t(8;21) or t(15;17)) or high risk myelodysplastic syndrome (MDS) (defined as bone marrow blasts > or = 5%) are eligible. Patients may be in remission at the time of entry.
3. Patients with adequate organ function and performance status criteria measured by:

   1. Karnofsky score greater than or equal to 70% or Performance status of < or = 2 by the Eastern Cooperative Oncology Group (ECOG) scale
   2. Adequate liver function (bilirubin of < 2mg/dL, serum glutamate pyruvate transaminase < 3 * ULN) and renal function (creatinine < 2mg/dL)
4. Signed informed consent indicating that patients are aware of the investigational nature of this study in accordance with the regulations of Loyola University Medical Center
5. Patients must have undergone allogeneic stem cell transplant within 40-60 days before starting treatment and be self-sufficient in caloric intake along with no active graft vs. host disease

Exclusion Criteria:

1. Nursing and pregnant females are excluded.
2. Active and uncontrolled infections will cause patients to be excluded.
3. Patients already receiving valproic acid or receiving other anticonvulsants will be excluded.
4. Low risk AML in complete remission 1, will not be candidates for this study.
5. Patients with an absolute neutrophil count less than 1500 will be excluded
6. Patients with platelets less than 50,000 will be excluded
7. Children less than 2 years of age will be excluded due to increased hepatotoxicity from valproic acid in this age group

Ages: 2 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
  Number of participants that survive post transplant for 1 year.

SECONDARY OUTCOMES:
Disease Relapse | Day 0 to the day of first recurrance
  The time to relapse is from Day 0 to the day of first hematologic, cytogenetic, or radiological evidence of recurrent disease.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stiff, MD, Principal Investigator — Faculty
Locations (1):
- Loyola University Cardinal Bernardin Cancer Center, Maywood, Illinois, United States